CLINICAL TRIAL: NCT01095497
Title: An Open-Label Multiple-Dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Subcutaneous (SC) Versus Intravenous (IV) Administration of CINRYZE in Adolescents and Adults With Hereditary Angioedema (HAE)
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Subcutaneous CINRYZE Administration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 0624-200; SPD616-200 (Other: Sponsor)
Record Dates: First submitted 2010-02-22; First posted 2010-03-30 (Estimated); Results first posted 2012-03-08 (Estimated); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Hereditary Angioedema
Keywords: HAE; C1 inhibitor (C1INH); Subcutaneous
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — SERPING1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV CINRYZE First, Then SC CINRYZE Dose 1 (Experimental)
  Interventions: Biological: CINRYZE
- IV CINRYZE First, Then SC CINRYZE Dose 2 (Experimental)
  Interventions: Biological: CINRYZE

INTERVENTIONS:
Biological: CINRYZE — C1 esterase inhibitor (human)

SUMMARY:
The objectives of the study are to:

1. Evaluate the safety and tolerability of CINRYZE administered by subcutaneous injection in subjects with hereditary angioedema
2. Characterize the pharmacokinetics and pharmacodynamics of CINRYZE administered by subcutaneous injection
3. Assess the immunogenicity of CINRYZE following subcutaneous administration

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this protocol, a subject must:

1. Have a confirmed diagnosis of HAE.
2. During the 3 consecutive months prior to screening, have a history of less than 1 HAE attack per month (average) treated with C1INH therapy or any other blood products, ecallantide (Kalbitor), icatibant (Firazyr), antifibrinolytics (e.g., tranexamic acid), IV fluids, or narcotic analgesics.
3. Agree to strictly adhere to the protocol-defined schedule of assessments and procedures.

Exclusion Criteria:

To be eligible for this protocol, a subject must not:

1. Have received C1INH therapy or any blood products for treatment or prevention of an HAE attack within 14 days prior to the first dose.
2. Have received any ecallantide (Kalbitor), icatibant (Firazyr), or antifibrinolytics (e.g., tranexamic acid) within 14 days prior to the first dose.
3. Have any change (start, stop, or change in dose) in androgen therapy (e.g., danazol, oxandrolone, stanozolol, testosterone) within 14 days prior to the first dose.
4. If female, have started taking or changed the dose of any hormonal contraceptive regimen or hormone replacement therapy (i.e., estrogen/progestin containing products) within 3 months prior to the first dose.
5. Have a history of abnormal blood clotting or other coagulopathy.
6. Have a history of allergic reaction to CINRYZE or other blood products.
7. Be pregnant or breastfeeding.
8. Have received an immunization within 30 days prior to the first dose.
9. Have participated in any other investigational drug study within 30 days prior to the first dose.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-06-07 (Actual); Primary Completion 2010-12-16 (Actual); Study Completion 2010-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (7):
- United States (7):
  - Allergy, Asthma and Immunology Associates, Scottsdale, Arizona
  - Allergy and Asthma Clinical Research, Inc., Walnut Creek, California
  - Family Allergy and Asthma Center, Atlanta, Georgia
  - Institute for Asthma and Allergy, Chevy Chase, Maryland
  - Allergy, Asthma and Dermatology Research Center, Lake Oswego, Oregon
  - AARA Research Center, Dallas, Texas
  - Marycliff Allergy Specialists, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- IV CINRYZE First, Then SC CINRYZE Dose 1: Subjects participated in two 18-day treatment periods, separated by a washout period of at least 14 days. In Period 1, subjects received 1000 Units of intravenous (IV) CINRYZE twice weekly for two weeks. In Period 2, subjects received 1000 Units of subcutaneous (SC) CINRYZE twice weekly for two weeks.
- IV CINRYZE First, Then SC CINRYZE Dose 2: Subjects participated in two 18-day treatment periods, separated by a washout period of at least 14 days. In Period 1, subjects received 1000 Units of IV CINRYZE twice weekly for two weeks. In Period 2, subjects received 2000 Units of SC CINRYZE twice weekly for two weeks.
Period: Intravenous CINRYZE
Arm/Group | IV CINRYZE First, Then SC CINRYZE Dose 1 | IV CINRYZE First, Then SC CINRYZE Dose 2
Started | 14 | 12
Completed | 13 | 12
Not Completed | 1 | 0
Period: Subcutaneous CINRYZE
Arm/Group | IV CINRYZE First, Then SC CINRYZE Dose 1 | IV CINRYZE First, Then SC CINRYZE Dose 2
Started | 13 | 12
Completed | 12 | 12
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- IV CINRYZE First, Then SC CINRYZE Dose 1: Subjects participated in two 18-day treatment periods, separated by a washout period of at least 14 days. In Period 1, subjects received 1000 Units of IV CINRYZE twice weekly for two weeks. In Period 2, subjects received 1000 Units of SC CINRYZE twice weekly for two weeks.
- Total: Total of all reporting groups
Arm/Group | IV CINRYZE First, Then SC CINRYZE Dose 1 | IV CINRYZE First, Then SC CINRYZE Dose 2 | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (12.70) | 37.3 (15.92) | 32.7 (14.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Adverse Events, Number of Subjects With Local Injection Site Reactions, and Number of Subjects Who Discontinue Study Drug or Withdraw From the Study.
Time Frame: 18 days in each treatment period
Population: Safety Analysis Set
Measure: Number; unit: Participants
Groups:
- Intravenous (IV) CINRYZE: 1000 Units of IV CINRYZE twice weekly for two weeks
- Subcutaneous (SC) CINRYZE Dose 1: 1000 Units of SC CINRYZE twice weekly for two weeks
- SC CINRYZE Dose 2: 2000 Units of SC CINRYZE twice weekly for two weeks
Arm/Group | Intravenous (IV) CINRYZE | Subcutaneous (SC) CINRYZE Dose 1 | SC CINRYZE Dose 2
Number analyzed (Participants) | 26 | 13 | 12
Participants
  Number of subjects with adverse events | 12 (0.019) | 10 (0.027) | 11 (0.010)
  Number of subjects with injection site reactions | 1 (0.033) | 10 (0.032) | 11 (0.010)
  Number of subjects who discontinued study drug | 1 | 0 | 0
  Number of subjects who withdrew from the study | 1 | 1 | 0

2. Secondary Outcome: Mean Change C1 Inhibitor (C1INH)
Description: Mean Change in Baseline in Observed Plasma Concentration of C1 Inhibitor (C1INH) Antigen. Baseline-corrected concentrations were derived by subtracting the observed pre-dose concentrations on Day 1 of each treatment period from each observed concentration.
Time Frame: 18 days in each treatment period
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- Intravenous (IV) CINRYZE: 1000 Units of IV CYNRYZE twice weekly for two weeks
- Subcutaneous (SC) CYNRYZE Dose 1: 1000 Units of SC CYNRYZE twice weekly for two weeks
- SC Dose 2: 2000 Units of SC CINRYZE twice weekly for two weeks
Arm/Group | Intravenous (IV) CINRYZE | Subcutaneous (SC) CYNRYZE Dose 1 | SC Dose 2
Number analyzed (Participants) | 25 | 13 | 12
g/L
  1 hour (h) post Dose 1 | 0.075 (0.023) | -0.002 (0.008) | -0.001 (0.006)
  2 h post Dose 1 | 0.070 (0.021) | -0.002 (0.008) | -0.001 (0.004)
  3 h post Dose 1 | 0.070 (0.023) | -0.002 (0.007) | -0.002 (0.007)
  4 h post Dose 1 | 0.065 (0.022) | 0.003 (0.005) | 0.003 (0.007)
  6 h post Dose 1 | 0.064 (0.018) | 0.002 (0.009) | 0.006 (0.007)
  8 h post Dose 1 | 0.062 (0.019) | 0.003 (0.010) | 0.009 (0.008)
  24 h post Dose 1 | 0.049 (0.016) | 0.016 (0.023) | 0.021 (0.011)
  48 h post Dose 1 | 0.035 (0.017) | 0.019 (0.030) | 0.028 (0.009)
  Pre-Dose 2 | 0.027 (0.024) | 0.011 (0.021) | 0.026 (0.008)
  1 h post Dose 2 | 0.088 (0.036) | 0.013 (0.022) | 0.027 (0.009)
  120 h post Dose 1 | 0.042 (0.018) | 0.024 (0.032) | 0.037 (0.009)
  Pre-Dose 3 | 0.019 (0.016) | 0.012 (0.024) | 0.024 (0.009)
  1 h post Dose 3 | 0.093 (0.028) | 0.012 (0.024) | 0.024 (0.010)
  Pre-Dose 4 | 0.024 (0.020) | 0.019 (0.034) | 0.030 (0.015)
  1 h post Dose 4 | 0.098 (0.035) | 0.010 (0.031) | 0.031 (0.012)
  2 h post Dose 4 | 0.092 (0.032) | 0.012 (0.028) | 0.029 (0.015)
  3 h post Dose 4 | 0.087 (0.031) | 0.014 (0.030) | 0.031 (0.014)
  4 h post Dose 4 | 0.086 (0.031) | 0.016 (0.029) | 0.035 (0.015)
  6 h post Dose 4 | 0.081 (0.031) | 0.016 (0.028) | 0.034 (0.015)
  8 h post Dose 4 | 0.080 (0.029) | 0.017 (0.032) | 0.036 (0.012)
  24 h post Dose 4 | 0.060 (0.025) | 0.026 (0.032) | 0.043 (0.009)
  48 h post Dose 4 | 0.038 (0.022) | 0.022 (0.028) | 0.045 (0.012)
  72 h post Dose 4 | 0.025 (0.022) | 0.017 (0.026) | 0.037 (0.013)
  120 h post Dose 4 | 0.008 (0.018) | 0.003 (0.022) | 0.025 (0.012)
  168 h post Dose 4 | 0.005 (0.016) | 0.005 (0.024) | 0.017 (0.011)

3. Secondary Outcome: Mean Change C4 Compliment
Description: Mean Change in Baseline in Observed Plasma Concentration of C4 Compliment. Baseline-corrected concentrations were derived by subtracting the observed pre-dose concentrations on Day 1 of each treatment period from each observed concentration.
Time Frame: 18 days in each treatment period
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Intravenous (IV) CINRYZE | Subcutaneous (SC) CYNRYZE Dose 1 | SC Dose 2
Number analyzed (Participants) | 25 | 13 | 12
mg/L
  1 hour (h) post Dose 1 | -7.5 (15.4) | -12.9 (15.6) | 0.1 (8.0)
  2 h post Dose 1 | -0.6 (10.2) | -3.8 (18.2) | -3.3 (8.9)
  3 h post Dose 1 | -1.3 (13.5) | -0.6 (10.9) | 2.5 (11.1)
  4 h post Dose 1 | 2.7 (14.8) | -5.3 (18.5) | 8.8 (23.7)
  6 h post Dose 1 | 12.0 (24.8) | -0.6 (37.1) | 8.1 (21.0)
  8 h post Dose 1 | 13.0 (20.7) | -8.2 (24.6) | 11.2 (27.4)
  24 h post Dose 1 | 25.5 (30.3) | 2.9 (25.4) | 14.3 (12.7)
  48 h post Dose 1 | 31.0 (25.3) | 6.2 (23.1) | 23.3 (18.0)
  Pre-Dose 2 | 29.5 (23.9) | 8.7 (23.4) | 30.2 (15.3)
  1 h post Dose 2 | 24.7 (26.4) | 5.6 (23.7) | 31.8 (19.3)
  120 h post Dose 1 | 53.1 (24.4) | 21.7 (22.7) | 37.9 (28.1)
  Pre-Dose 3 | 28.1 (29.3) | 7.3 (20.6) | 57.3 (46.6)
  1 h post Dose 3 | 26.0 (20.9) | 5.8 (22.3) | 40.4 (26.5)
  Pre-Dose 4 | 34.4 (26.9) | 5.4 (27.6) | 50.5 (18.7)
  1 h post Dose 4 | 28.6 (27.0) | 1.9 (25.0) | 51.2 (22.6)
  2 h post Dose 4 | 29.4 (26.2) | 6.6 (25.2) | 49.4 (21.1)
  3 h post Dose 4 | 34.7 (24.9) | 8.8 (25.0) | 54.9 (26.4)
  4 h post Dose 4 | 33.7 (31.1) | 9.2 (27.0) | 62.8 (41.2)
  6 h post Dose 4 | 39.4 (26.8) | 4.2 (26.5) | 67.1 (57.3)
  8 h post Dose 4 | 41.9 (30.1) | 6.4 (27.8) | 67.3 (53.4)
  24 h post Dose 4 | 56.5 (36.0) | 4.0 (23.8) | 49.3 (31.6)
  48 h post Dose 4 | 54.9 (34.6) | 8.2 (23.6) | 56.5 (29.2)
  72 h post Dose 4 | 46.1 (36.2) | 10.9 (27.9) | 62.6 (43.8)
  120 h post Dose 4 | 11.0 (32.1) | -4.5 (26.0) | 47.2 (32.3)
  168 h post Dose 4 | -0.6 (27.1) | 2.2 (24.5) | 36.5 (32.9)

4. Secondary Outcome: Number of Participants With C1 Inhibitor (INH) Antibodies
Time Frame: 18 days in each treatment period
Measure: Number; unit: Participants
Arm/Group | Intravenous (IV) CINRYZE | Subcutaneous (SC) CINRYZE Dose 1 | SC CINRYZE Dose 2
Number analyzed (Participants) | 26 | 13 | 12
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Intravenous (IV) CINRYZE | Subcutaneous (SC) CINRYZE Dose 1 | SC CINRYZE Dose 2
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 8/26 | 10/13 | 11/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intravenous (IV) CINRYZE (N=26) | Subcutaneous (SC) CINRYZE Dose 1 (N=13) | SC CINRYZE Dose 2 (N=12)
Injection site pain (General disorders) | 0 | 10 | 8 — 39% mild, 51% moderate, 10% severe
Hereditary angioedema (Congenital, familial and genetic disorders) | 5 | 2 | 0 — 64% mild, 27% moderate, 9% severe
Injection site erythema (General disorders) | 0 | 4 | 2 — 75% mild, 25% moderate
Headache (Nervous system disorders) | 1 | 1 | 2 — 25% mild, 75% moderate
Injection site hematoma (General disorders) | 0 | 1 | 2 — 100% mild
Injection site pruritus (General disorders) | 0 | 2 | 1 — 100% mild
Acne cystic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 — 50% mild, 50% moderate
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0 — 50% mild, 50% moderate
Injection site swelling (General disorders) | 0 | 1 | 1 — 100% mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement. Most restrictive provision - PI will not publish results until after first of: multicenter publication is published or 24 months from study end. Thereafter, PI may publish his results. PI must provide copy of proposed publication to Sponsor for pre-review. If Sponsor requests, PI must delete Sponsor confidential information before publication and/or delay publication for 60 days so Sponsor can file for patents or take other action to protect its patent rights.